CLINICAL TRIAL: NCT06480747
Title: The Effects of Strength Training on Neuromuscular Function and Muscle Lipids.
Brief Title: Strength Training and Muscle Lipids
Acronym: Strength-Lip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Strength and Conditioning Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00160469
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: exercise; muscle cross-sectional area; intramyocellular lipids; extramyocellular lipids; muscle power; motor unit
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise training (Experimental)
  Interventions: Other: Resistance exercise training
- Control (No Intervention)

INTERVENTIONS:
Other: Resistance exercise training — Participants will strength train via linear periodization resistance exercise training.
  Arms: Resistance exercise training

SUMMARY:
The purpose of this study is examine the effects of 8 weeks (3 days/week) of resistance exercise training in children 8 to 10 years of age on muscle strength and power, motor unit activation, and lipid profiles of the vastus lateralis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer males and females ages 8 - 10 years.

Exclusion Criteria:

* No history or ongoing neuromuscular diseases.
* No history or ongoing musculoskeletal injuries.
* No history or ongoing disease that effects metabolism.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Change in muscular power of the leg extensors, as measured with isokinetic strength testing. | Baseline, following the intervention (9 weeks)
  The score will reflect the muscular power of the leg extensors. The higher score, reflects greater muscular strength.

SECONDARY OUTCOMES:
Change from baseline in thigh muscle cross-sectional area | Baseline, following the intervention (9 weeks)
  Scores are measured cross-sectional area from ultrasound images. The higher score, reflects greater muscle size of the leg extensors.

OTHER OUTCOMES:
Change from baseline in intramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a concentration. The higher score, reflects more fat in the fibers.
Change from baseline in extramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a concentration. The higher score, reflects more fat in the fibers.
Change from baseline in the fatty acid saturation levels of the extramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a saturation level of fatty acids in the extramyocellular lipid. The higher score, reflects greater fatty acid saturation.
Change from baseline in the fatty acid saturation levels of the intramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a saturation level of fatty acids in the intramyocellular lipid. The higher score, reflects greater fatty acid saturation.
Change from baseline in motor unit activation, as measured with surface electromyography decomposition. | baseline, following the intervention (9 weeks)
  The score will reflect the firing rates of recorded motor units. The higher score, reflects greater motor unit activation.
Change in total body lean mass, as measured with bioelectrical impedance analysis. | baseline, following the intervention (9 weeks)
  The score will reflect the lean mass. The higher score, reflects greater lean mass.
Change in total body fat mass, as measured with bioelectrical impedance analysis. | baseline, following the intervention (9 weeks)
  The score will reflect the fat mass. The higher score, reflects greater fat mass.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hoglund Biomedical Imaging Center, Kansas City, Kansas
  - Neuromechanics Laboratory, Lawrence, Kansas
  - Exercise and Human Performance Laboratory, Overland Park, Kansas
  - Metabolic and Body Composition Laboratory, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No